CLINICAL TRIAL: NCT03955640
Title: A Pilot Trial of Hyperthermia in Combination With Olaparib in Breast Cancer Patients With Chest Wall Recurrences
Brief Title: Hyperthermia and Olaparib in Treating Breast Cancer Patients With Chest Wall Recurrences
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI decided not to move forward because of low accrual
Sponsor: Thomas Jefferson University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19P.117; JT 13333 (Other: JeffTrial Number)
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Malignant Neoplasm in the Chest Wall; Recurrent Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — olaparib; Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (olaparib, hyperthermia) (Experimental): Patients receive olaparib PO BID. Treatment continues for 4 weeks in the absence of disease progression and unacceptable toxicity. Beginning week 2, patients also undergo hyperthermia treatment over 1 hour twice weekly for 3 weeks in the absence of disease progression and unacceptable toxicity.
  Interventions: Drug: Olaparib; Procedure: Hyperthermia Treatment; Other: Questionnaire Administration; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Olaparib — Given PO
  Other Names: 763113-22-0; AZD2281; KU-0059436; Lynparza; PARP Inhibitor AZD2281
Procedure: Hyperthermia Treatment — Undergo hyperthermia treatment
  Other Names: Clinical Hyperthermia; Diathermy; Hyperthermia; hyperthermia therapy
Other: Questionnaire Administration — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase I trial studies the side effects and best dose of olaparib when given with hyperthermia in treating patients with breast cancer that has come back in the chest wall. Olaparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Hyperthermia treatment may kill or damage tumor cells by heating them to several degrees above normal body temperature. Giving olaparib and hyperthermia treatment may work better in treating patients with breast cancer that has come back in the chest well compared to standard of care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the dose limiting toxicities and maximum tolerated dose of olaparib given in combination with chest wall hyperthermia in patients with locally advanced or metastatic breast cancer with chest wall recurrences who have wild-type BRCA status (patients with germline BRCA mutations are excluded from this study).

SECONDARY OBJECTIVES:

I. To determine the local progression free survival (in months) for patients with chest wall recurrences defined as time to progression of disease on chest wall with olaparib with hyperthermia.

II. To determine the 1-year progression free survival (in months) for patients with chest wall recurrences treated with olaparib with hyperthermia.

III. To determine the best local overall response rate of chest wall after the combination of hyperthermia and olaparib.

IV. To determine the quality of life and pain scores before, during and after treatment as measured by the Edmonton Symptom Assessment System which includes a pain score and 8 other subjective measures of wellness for cancer patients (0 to 10).

EXPLORATORY OBJECTIVES:

I. To evaluate BRCA1/2 levels by immunohistochemistry and explore if hyperthermia induced BRCA1/2 expression.

II. To evaluate HR (homologous recombination) competency by RAD51 foci and explore if hyperthermia induces homologous recombination in breast tissue.

III. To explore deoxyribonucleic acid (DNA) damage as measured by gammaH2AX and comet assay in cells dissociated from biopsy tissues.

OUTLINE: This is a dose-escalation study of olaparib.

Patients receive olaparib orally (PO) twice daily (BID). Treatment continues for 4 weeks in the absence of disease progression and unacceptable toxicity. Beginning week 2, patients also undergo hyperthermia treatment over 1 hour twice weekly for 3 weeks in the absence of disease progression and unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients regardless of estrogen receptor (ER)/progesterone receptor (PR)/HER2 status and have breast cancer recurrence on the chest wall
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol
* Provision of signed and dated, written informed consent form prior to any mandatory study specific procedures, sampling, and analyses
* Hemoglobin >= 10.0 g/dL with no blood transfusion in the past 28 days (within 28 days prior to administration of study treatment)
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (measured within 28 days prior administration of study treatment)
* Platelet count >= 100 x 10^9/L (measured within 28 days prior to administration of study treatment)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (measured within 28 days prior to administration of study treatment)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) / alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal unless liver metastases are present in which case they must be =< 5x ULN (measured within 28 days prior to administration of study treatment)
* Patients must have creatinine clearance estimated of >= 51 mL/min using the Cockcroft-Gault equation or based on a 24 hour urine test (measured within 28 days prior to administration of study treatment)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Patients must have a life expectancy >= 16 weeks
* Breast cancer with chest wall disease that is at least 2 cm in size at the greatest dimension
* Patients will be eligible for this trial regardless of number of lines of therapy and after adjuvant chemotherapy with recurrence on the chest wall
* Patients with hormone receptor positive disease who discontinue endocrine therapy two weeks prior to initiating study treatment are eligible
* Body mass index (BMI): 15 to 50 at the time of consent
* Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of initiating study treatment and confirmed prior to treatment on day 1 and willingness to use effective contraception during study treatment and for at least 30 days after last dose of study drug. Postmenopausal is defined as:

  * Amenorrhea for 1 year or more following cessation of exogenous hormonal treatments
  * Luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels in the post menopausal range for women under 50
  * Radiation-induced oophorectomy with last menses > 1 year ago
  * Chemotherapy-induced menopause with > 1 year interval since last menses
  * Surgical sterilization (bilateral oophorectomy or hysterectomy)

Exclusion Criteria:

* As judged by the investigator, any evidence of non-compliance which in the investigator's opinion makes it undesirable for the patient to participate in the trial
* Patients with rapidly progressing disease
* Metastatic disease should not be progressing so as to require systemic treatment within 4 weeks of enrollment based on clinical assessment by the investigator
* Metastatic disease should not be progressing so as to require palliative treatment within 4 weeks of enrollment based on clinical assessment by the investigator
* Other malignancy unless curatively treated with no evidence of disease for >= 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), stage 1, grade 1 endometrial carcinoma
* Resting electrocardiogram (EKG) indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g. unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, corrected QT interval by Fridericia [QTcF] prolongation > 500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome
* Persistent toxicities caused by previous cancer therapy >= grade 2, excluding alopecia and neuropathy
* Patients with current or previous diagnosis of myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML)
* Patients with symptomatic uncontrolled brain metastases or spinal cord metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on high resolution computed tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication
* Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV)
* Any previous treatment with PARP inhibitor, including olaparib
* Subjects with a known hypersensitivity to olaparib or any of the excipients of the product
* Patients with a known hypersensitivity to hyperthermia
* Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment
* Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks
* Concomitant use of known strong CYP3A inducers (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's wort) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents
* Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of surgery
* Patients with known active hepatitis B or C
* Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable outside of 28 days prior to enrollment)
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
* Any patient with a known germline BRCA1 or 2 mutation
* Participation in another clinical study with an investigational product administered in the last 2 months
* Previous enrollment in the present study
* Breast feeding women
* Involvement in the planning and/or conduct of the study
* No radiotherapy, treatment with cytotoxic agents, biologic agents within 3 weeks prior to beginning treatment on this study. Patients must have recovered from the acute toxicities of any prior treatment with cytotoxic drugs to =< grade 1 (allowance for grade 2 alopecia and neuropathy) in order to be eligible. Patients who underwent post-mastectomy radiation will not be excluded from this study

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2021-08-26 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 1 year post treatment
  Will be continually assessed according to the National Cancer Institute Common Toxicity Criteria for Adverse Advents (CTCAE version [v]5.0).

SECONDARY OUTCOMES:
Local progression free-survival (PFS) | From first dose of olaparib to the date of the first documented disease progression or recurrence on the chest wall, assessed up to 1 year
  Will be reported as Kaplan-Meier survival curves with the median survival time with 95% confidence interval. Will be analyzed using log-rank test as well as Cox proportional hazard models.
PFS | From first dose of olaparib to the date of the first documented disease progression or recurrence, or death due to any cause, whichever occurs first, assessed up to 1 year
  Will be assessed using Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Will be reported as Kaplan-Meier survival curves with the median survival time with 95% confidence interval. Will be analyzed using log-rank test as well as Cox proportional hazard models.
Best local overall response rate (ORR) | Up to 1 year post treatment
  Defined as the number of subjects with a best overall response (BOR) defined as a complete response (CR) or partial response (PR) divided by the number of enrolled subjects. The proportion of patients will be summarized together with the appropriate 95% confidence interval. The binary endpoint of ORR will be compared by test on proportions.
Quality of life (QOL) | Up to 1 year post treatment
  Defined by the Edmonton Symptom Assessment System (ESAS) using nine subjective patient measures of well-being including pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, well-being, shortness of breath. These will be rated by the patients during each visit (visits 1-6) and the change in values will correlate to an improvement in quality of life (a positive change will correlate to an improvement and a negative change will correlate to a worsening of pain). The multinominal/ordinal endpoints in QOLs will be summarized in frequencies ad proportions and compared using trend test.
Pain scores | Up to 1 year post treatment
  Defined by the Edmonton Symptom Assessment System (ESAS) using nine subjective patient measures of well-being including pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, well-being, shortness of breath. These will be rated by the patients during each visit (visits 1-6) and the change in values will correlate to an improvement in quality of life (a positive change will correlate to an improvement and a negative change will correlate to a worsening of pain).

OTHER OUTCOMES:
BRCA1/2 expression patterns | Up to 1 year post treatment
  The proportion of patients with BRCA1/2 positive tumors among the patients by immunohistochemistry (IHC) will be estimated along with appropriate 95% confidence intervals. Similarly, the proportion of samples where BRCA1/2 status can successfully be obtained will be estimated as a measure of feasibility. Finally, the proportion of samples in which BRCA1/2 status is altered upon treatment will be estimated along with the appropriate 95% confidence intervals.
Homologous recombination (HR) capacity | Up to 1 year post treatment
  Analysis of tumor explant data and the assessment of HR capacity will use linear or generalized linear mixed effects models for repeated measurements depending on the outcome of interest.
Deoxyribonucleic acid (DNA) damage | Up to 1 year post treatment
  Analysis of tumor explant data and the assessment of DNA damage will use linear or generalized linear mixed effects models for repeated measurements depending on the outcome of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Maysa Abu-Khalaf, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States